CLINICAL TRIAL: NCT03675269
Title: Adjunctive Hyperbaric Oxygen Therapy (HBOT) for Lower Extermity Diabetic Ulcer: A Prospective Double-Blind, Randomized Control Clinical Trail
Brief Title: Adjunctive Hyperbaric Oxygen Therapy (HBOT) for Lower Extermity Diabetic Ulcer:
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was moved to another location with involvement of different researchers
Sponsor: King Hamad University Hospital, Bahrain (Other)
Collaborators: University of Stellenbosch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KingHamadUHBahrain
Record Dates: First submitted 2018-08-27; First posted 2018-09-18 (Actual); Last update posted 2019-02-28 (Actual); Status verified 2019-02

CONDITIONS: Ulcer Foot; Diabetic Foot Ulcer
MeSH Terms: conditions — Foot Ulcer; Diabetic Foot

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): HBOT
  Interventions: Other: HBOT; Behavioral: Standard wound care
- Control (Active Comparator): Standard wound care
  Interventions: Behavioral: Standard wound care

INTERVENTIONS:
Other: HBOT — Standard practice
  Arms: Treatment
Behavioral: Standard wound care — Standard wound care

SUMMARY:
Diabetic foot ulcers are associated with high risk of amputation. About 50% of patients undergoing non-traumatic lower limb amputations are diabetics5. The 5-year amputation rate is estimated to be 19% with a mean time to amputation 58 months since the onset of an diabetic foot ulcer6.Because infection and tissue hypoxia are the major contributing factors for non-healing diabetic foot ulcers, hyperbaric oxygen therapy (HBO) carries a potential benefit for treating these problematic wounds that do not respond to standard therapy.

The role of oxygen in the wound healing cascade and subsequent combatting action against bacterial invasion, especially anaerobes, is well documented.14 Delayed or arrested healing and the development of infection is a direct result from decreased perfusion and poor oxygenation of tissue.15 The presence of wound hypoxia is an major etiological pathway in the development of chronic non-healing diabetic foot ulcers

DETAILED DESCRIPTION:
1 KHUH Research Center

The Premise of the study:

Hyperbaric Oxygen as adjunctive therapy is effective towards the healing of diabetic lower extremity ulcers and has a role to play in major amputation prevention for persons with Diabetes Mellitus.

Title of the project:

Adjunctive Hyperbaric Oxygen Therapy (HBOT) for Lower Extremity Diabetic Ulcers: A Prospective, Double-Blind, Randomized, Controlled Clinical Trial Background Diabetes Mellitus is a major health problem with significant morbidity and mortality. The number of people with diabetes mellitus worldwide is estimated at 285 million in 2010; and expected to increase to 438 million by 20301. In western countries, like the United Kingdom, diabetic foot ulcers are the most commonly found chronic wound2. A diabetic foot ulcer is defined as a 'full thickness' lesion of the skin, that is, a wound penetrating through the dermis below the ankle joint3. The lifetime risk of developing foot ulcers in diabetics is estimated to be 15%4. These ulcers may heal with proper wound care, but some may become chronic and others may lead to amputation. These different outcomes are influenced by several risk factors including, among others, peripheral arterial disease (ischemia), peripheral neuropathy, mechanical foot deformity, poor foot care and inappropriate shoe wear.

Diabetic foot ulcers are associated with high risk of amputation. About 50% of patients undergoing non-traumatic lower limb amputations are diabetics5. The 5-year amputation rate is estimated to be 19% with a mean time to amputation 58 months since the onset of an diabetic foot ulcer6.Because infection and tissue hypoxia are the major contributing factors for non-healing diabetic foot ulcers, hyperbaric oxygen therapy (HBO) carries a potential benefit for treating these problematic wounds that do not respond to standard therapy7.

Vascular: Approximately 35% of diabetic foot ulcers result from peripheral vasculopathy with an additional 15-20% caused by mixed neuropathic-vasculopathic pathology8. There is an accelerated development of atherosclerosis in the distal arteries (tibial and peroneal arteries) of diabetic patients with the dorsalis pedis artery often spared. Abnormal smooth muscle tone and decreased perfusion exacerbate these changes. On a macrovascular level, thickening of the basement membrane and abnormal endothelial function is often found. Tissue ischemia may be worsened by capillary thrombosis and by impaired neurogenic control.9 The microcirculation of diabetic patients exhibits characteristic structural changes such as the reduction in the size of capillaries and thickening in basement membrane that impairs the normal hyperemic or vasodilatory response to injury10, 11 and interferes with transportation of nutrients and oxygen. Arterial thrombosis commonly develops in the presence of pre-existing atherosclerotic 2 changes in the vascular endothelium, as a result of low blood flow and increased blood viscosity or a pro-coagulative state. All of these changes are exacerbated by a smoking habit (cigarettes, cigars or water pipes) by inducing peripheral vasoconstriction that reduces available oxygen to tissue by 20-30% per cigarette for one hour.12 It induces alterations in lipid metabolism, increases platelet aggregation, and increase blood viscosity.12 Pressure: Peripheral neuropathy is the most common cause of foot ulcers and is present in 78% of the ulcer formation pathway.8 Foot deformity is the most common underlying cause and that is leading to unequal pressure redistribution and subsequent ulceration. Poor glycemic control and poor glycemic control increase the risk of neuropathy and is directly linked to the duration of living with diabetes (>15 years carrying a higher risk for developing neuropathy13), manifesting in all three components of the nervous system (autonomic, motor and sensory).

Autonomic neuropathy of the foot results in loss of sweat and oil gland function leading to dry cracked skin prone to bacterial infections; the loss of sympathetic vascular tone that leads to vasodilatation and the development of edema8.

Motor neuropathy causes loss of nerve supply to the intrinsic foot muscles with subsequent imbalance of the long flexor and extensor tendons. This produces an anatomic foot deformity with hyperextension of the toes, dropdown of the metatarsal heads and distal movement of the protective fat pad leading to pressure imbalance, callus formation and underlying skin breakdown.

In sensory neuropathy the loss of the protective components of the foot is rendering patients unaware of repeated traumas and small injury as a pain response is absent. A wound remain undetected, worsen, becomes secondarily infected with the patient usually late in presenting to formal health care, adding to the severity of the foot condition on assessment.

The role of oxygen in the wound healing cascade and subsequent combatting action against bacterial invasion, especially anaerobes, is well documented.14 Delayed or arrested healing and the development of infection is a direct result from decreased perfusion and poor oxygenation of tissue.15 The presence of wound hypoxia is an major etiological pathway in the development of chronic non-healing diabetic foot ulcers.16

Measurement of tissue oxygenation is done with transcutaneous oximetry (TcPO2) and provides a simple, noninvasive diagnostic technique for an objective assessment of local tissue perfusion and oxygenation.17 TcPO2 measurements are frequently used in the assessment of diabetic ulcers to:

1. Assess the severity of tissue hypoxia;
2. Determine a saturation response to 100% oxygen;
3. Serve as a predictor for response to HBO therapy;
4. Provide a guideline on when to stop therapy; and
5. Define healable levels for lower limb amputation18. Studies have shown that an achieved value below 40 mmHg on breathing normal air, is associated with poor healing of diabetic foot ulcers adding to amputation risk, while values higher than 40 mmHg is likely to yield spontaneous resolution of foot ulcers.19 Saturated TcPO2 values (breathing 100% oxygen via a non-rebreather mask for 15 minutes) that exceeds a cutoff value of 200 mmHg, is associated with a positive predictive value to the extent of 74% for wound healing improvement, or limb salvage following a therapeutic course of hyperbaric oxygen therapy.20 Level 1A evidence of the beneficial effect of HBO therapy on diabetic foot outcomes was initially scant with only two prospective RCT studies available before 2000.21, 22 One study was added in 200323 and 3 then a gap existed that was only filled in 201324 due to the difficulties associated with a trial using HBO as adjunctive modality. All of these studies have shown efficacy of HBO with the systematic review from Liu et al in 201325 showing a reduction of major limb amputations (minor amputations though present) and establishing a foundation for wound healing to progress (neovascularization and granulation stimulation). The retrospective cohort study of Margolis et al26 though, has disproved the effectiveness of HBO as modality in management of diabetic foot ulcers. Major limitations were identified on doing a systematic critique27 of that study with design, sample selection with inappropriate inclusions, unequal study arms, statistical usage of a propensity score to adjust for wound severity and unclear expected endpoints the most prevalent. This study has highlighted the difference between effectiveness (if something has been beneficially employed in the day to day setting) and efficacy (does it work) and that is the answer would like to provide with an effectiveness study in a prospective, rather than retrospective design.

Objectives of the study:

Study aim and objectives The aim of this study is to determine the effectiveness of 30 sessions of adjunctive hyperbaric oxygen therapy on the healing rate of diabetic lower extremity ulcers.

Primary objectives:

To compare between the treatment and control group:

The reduction of wound size at 4 weeks (granulation formation) as measured by the Silhouette three dimensional photography Time to achieve 80% wound surface reduction as measured by the Silhouette trajectory Time to achieve bipedal ambulation on an offloading device crossing the ankle joint The level of neovascularization achieved as measured by transcutaneous oximetry The proportion of patients ending up with a below knee amputation.

Secondary objectives:

Determine the TCpO2 criteria by which treatment response could be measured.Determine the TCpO2 criteria by which optimal treatment is assessed (to indicate completion of therapy).

Evaluate the role of minor amputations (one or more toes up to the mid foot) in saving the major limb (integrity of the knee and ankle joint) Evaluate the role of HBO in resolution of infection/osteomyelitis in conjunction with appropriate systemic antibiotics.

To determine and describe the side-effects of HBO therapy. 4 Improvement of quality of life with particular attention to pain. Setting: The hyperbaric and wound care unit of King Hamad University hospital, Kingdom of Bahrain

Design: A parallel prospective double-blind randomized placebo-controlled trial.

Sample size: 100-120 patients equally divided between the two treatment arms Sampling technique: Randomization by sealed envelope method to either Arm A or Arm B, both blinded to all apart from the primary researcher.

Timeframe of the study: 12-24 months in order to fill the appropriate sample size on an 80% confidence interval

Data Collection methods, instruments used and measurements:

1. Transcutaneous oxygen measurements on air and saturated values pre-treatment, 10 sessions, 20 sessions and 30 sessions
2. Silhouette 3 dimensional wound surface photography on each dressing change to determine % wound size reduction and create a healing trajectory in a quantifiable manner
3. Standard battery of HBO investigations pre-HBO: CBC, CXR, Foot x-ray, HbA1c, BMI
4. Daily pre- and post HBO chamber investigations: Vital signs, random blood glucose, Pain scale 5

Data management and analysis plan:

1. Basic descriptive statistics to describe the sample demographics and randomization achieved
2. T-test with Chi-square with confidence interval for healing achieved
3. Logistic regression with linear markers for neovascularization achieved
4. Analysis of co-variants for influence of confounding factors.

ELIGIBILITY:
Inclusion Criteria:

1. Any gender aged > 18 years.
2. Confirmed type 1 or type 2 Diabetes Mellitus patient, currently on anti-diabetic medication
3. Participant is to have at least one wound, which meets ALL of the following criteria: a. The ulcer to be present on the lower extremity below the ankle joint to make this study comparable to others done on diabetic patients b. Documented proof of chronicity (present for more than 3 months, despite conventional wound care).

   c. Wagner classification Grade 3 or higher as recommended by the Undersea and Hyperbaric Medical Society.
4. Meeting the selection for HBO criteria as determined by transcutaneous oxygen measurements.
5. Willing and able to provide an informed consent for the study and related procedures.

Exclusion Criteria:

1. Lower extremity or foot ulcers of non-diabetic peripheral vascular disease, venous, lymphedematous or neoplastic etiology.
2. Having any condition or previous treatment that is known to be a contra-indicated for hyperbaric oxygen therapy.
3. Pregnant or lactating females.
4. Candidate with proven macro-vascular compromise who is not eligible for vascular intervention surgery.
5. Previous treatment with hyperbaric oxygen therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-09-05 (Actual); Primary Completion 2019-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Change in wound size | 4 years
  The change of wound size at 4 weeks (granulation formation) as measured by the Silhouette three dimensional photography